CLINICAL TRIAL: NCT02767622
Title: Reversibility of Minimal Hepatic Encephalopathy Following Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Abdelhakam, Assistant Professor, Ain Shams University
Other Study IDs: 875
Record Dates: First submitted 2016-05-07; First posted 2016-05-10 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Minimal Hepatic Encephalopathy
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patient Group: Twenty right handed patients with biopsy-proven liver cirrhosis listed for liver transplantation.
  Interventions: Procedure: Liver transplantation
- Control Group: Twenty age-matched healthy persons. They were similar to the patient group in respect to the number of education years, sex, and handedness.

INTERVENTIONS:
Procedure: Liver transplantation
  Groups: Patient Group

SUMMARY:
This study included 20 patients listed for liver transplantation in addition to 20 age- and sex- matched controls. Neurological, psychiatric, laboratory and radiological examinations were performed for both patients and controls before and 6 months after liver transplantation. Assessment of cognitive functions by Trail Making Test A (TMT A), TMT B, Digit Symbol Test (DST), and Serial Dotting Test (SDT) was done before and after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Right handed patients with biopsy-proven liver cirrhosis listed for liver transplantation

Exclusion Criteria:

* Overt hepatic encephalopathy.
* Significant cortical atrophy or other structural brain changes revealed by conventional neuro-imaging.
* Regular use of psychotropic drugs, such as benzodiazepines.
* Known major psychiatric disorder.
* Less than 6 months of complete alcohol abstinence.
* Post-transplant toxic levels of immunosuppressive drugs.
* Patients unable to perform the tests (Illiterate or upper limb motor handicaps).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty right handed patients with biopsy-proven liver cirrhosis listed for liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Improvement of Psychometric tests. | 6 months following liver transplantation.

SECONDARY OUTCOMES:
Improvement of liver functions and MELD score following liver transplantation. | 6 months following liver transplantation.